CLINICAL TRIAL: NCT04849442
Title: Association of Jaw Dysfunction With Neck Disability in Subjects With Chronic Cervical Spine Disorders: An Observational Study
Brief Title: Association of Jaw Dysfunction With Neck Disability in Subjects With Chronic Cervical Spine Disorders
Status: Completed | Type: Observational
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, Mohamed Salah El-Sayed, Principal Investigator, Horus University
Other Study IDs: msalah_bfpt
Record Dates: First submitted 2021-04-10; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Musculoskeletal Pain; TMJ Pain; Cervical Pain
MeSH Terms: conditions — Musculoskeletal Pain; Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since TMJ and cervical pain incidence are rising and both structures are highly interrelated anatomically and functionally. And yet no standard protocol for TMD therapy The objective of this study is to state if there is a correlation between TMD and cervical dysfunction. To help reach a better diagnosis and a more holistic treatment. Forty volunteers (15 male and 25 female) between the ages of 20 to 40 were recruited. Cervical ROM was measured in all directions (rotation, flexion and extension, and sidebending) by CROM device, and a 10 cm plastic ruler marked in both centimeters and millimeters was used to measure TMJ vertical opening.

DETAILED DESCRIPTION:
Background: The incidence of temporomandibular dysfunction has been rapidly increasing in the past years especially among women and still no definite treatment protocol and that's due to the inter lapping of anatomy and neurology of this joint with other structures all over the body. The cervical spine dysfunction has a high incidence as well, and they are common to coexist as they are highly interrelated. Objective: The objective of this study is to emphasize the interrelation between cervical dysfunction and TMJ dysfunction by examining the relationship between cervical spine ROM and TMJ vertical opening ROM to provide better recognition of the etiology of TMJ dysfunction thus a holistic intervention. Materials and methods: It is a bivariate correlational research design. Forty subjects between the age of 20 -40 years (15male/ 25females) were recruited. Cervical ROM was measured by CROM device for all 6 cervical movements. The TMJ vertical mouth opening was measured by a 10 cm ruler. The CROM will be used consistent with standard clinical procedures, with 3 takes for each measurement to decrease human error. The measurements were taken one shot.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 20 and 40
2. Female and Male
3. Suffering from a reduced cervical ROM
4. No reported TMJ pain

   Exclusion Criteria:
   * 1) Tumor (anywhere in the body)
5. Recent trauma to the neck, torso or upper limb
6. Active inflammation in the cervical region, upper thoraxic spine and chest or upper limb
7. Recent use of orthodontics prostheses

Ages: 20 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: The patients included in this study were recruited at the outpatient clinic of physical therapy and El Kasr El Einy Hospital from June 2019 till August 2019. The standard procedure is that patients fill out an admission form and undergo an intake assessment. After examination, the patient, who had a cervical dysfunction, was asked if they would be willing to undergo an assessment for this study. Forty volunteers (15 male and 25 female) between the ages of 20 to 40 (mean 27.05 +- 3.93 )
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Cervical spine range of motion by CROM | "through study completion, an average of 3 months"
  measuring the change of cervical range of motion in all directions (rotation, flexion and extension, and side bending)

SECONDARY OUTCOMES:
TMJ vertical opening | "through study completion, an average of 3 months"
  measuring the change of TMJ vertical opening by the second device used was a 10 cm plastic ruler marked in both centimeters and millimeters was used in the measurements, with (ICC 2,K) varied from 0.90 to 1.0, placed between the upper and lower edges of the central incisors

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed El-Sayed, Assistant lecturer, Principal Investigator — Horus University in Egypt
Locations (1):
- Outpatient clinic, Faculty of Physical Therapy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No